CLINICAL TRIAL: NCT03955718
Title: Developing and Testing Motherly: An Automated Gamified Smartphone Application to Promote Mothers' Mental Health
Brief Title: Developing and Testing Motherly App: a Smartphone Application to Promote Mothers' Mental Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped because of delays in the development of the smartphone app intervention
Sponsor: University of Sao Paulo (Other)
Collaborators: Grand Challenges Canada (Other); Fundação Maria Cecilia Souto Vidigal (Other)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SB-POC-1810-20573
Record Dates: First submitted 2019-01-28; First posted 2019-05-20 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Maternal Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motherly App (Experimental): A smartphone app with an automated intervention that provides strategies to prevent maternal depression and to promote child development: (1) behavioral activation, (2) sleep hygiene, (3) physical activity, (4) social support, (5) nutrition, (6) prenatal care schedule, and (7) educational content.
  Interventions: Behavioral: Motherly App
- Educational App (Active Control) (Active Comparator): An app with educational content about gestation, maternal health and mental health, child development, etc.
  Interventions: Behavioral: Educational App (Active Control)

INTERVENTIONS:
Behavioral: Motherly App — The Motherly app is a behavioral intervention aimed at preventing maternal depression and promoting child development.
  Arms: Motherly App
Behavioral: Educational App (Active Control) — An app with educational content about gestation, maternal health and mental health, child development, etc.
  Arms: Educational App (Active Control)

SUMMARY:
The investigators plan to develop and test Motherly, a smartphone app to promote maternal mental health and child development. The Motherly app is visually appealing aimed at engaging the user with a minimalistic layout. The app will offer a gamified experience ideal for engaging youth in behaviors that can promote mental health, such as stimulating pleasure, productivity, and physical activities, connecting with peers, and eating healthy food. Pregnant women aged 16-34 living in Brazil will participate in the clinical trial to test the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Literate women in the first or second trimester of pregnancy
* Living in Brazil
* Owning a functional smartphone for personal use with Android or iOS operational system

Exclusion Criteria:

* High-risk pregnancy

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-25 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Maternal depression | At 3 months of the child's age
  Maternal depression measured by the Patient Health Questionnaire (PHQ-9), less than 10 points in the scale

SECONDARY OUTCOMES:
Quality of sleep: Bergen Insomnia Scale | Monthly up to 3 months of the child's age
  Quality of sleep measured by the Bergen Insomnia Scale
Quality of maternal diet: questionnaire | Monthly up to 3 months of the child's age
  Quality of maternal diet measured by a 14-item questionnaire developed for the present study.
Physical activity | Monthly up to 3 months of the child's age
  Physical activity measured by accelerator data from the smartphone.
Psychological well-being | Monthly up to 3 months of the child's age
  Psychological well-being measured by the Ryff's Psychological well-being scales
General well-being | 3 months of the child's age
  WHO-5 Well-Being Index
Maternal anxiety | 3 months of the child's age
  Maternal anxiety measured by the General Anxiety Disorder 7 scale
Maternal self-efficacy: General Self-efficacy Scale | 3 months of the child's age
  Maternal self-efficacy measured by the General Self-efficacy Scale
Quality of stimulation and support available to the child in the home environment: Home Observation for Measurement of the Environment | 3 months of the child's age
  Quality of stimulation and support available to the child in the home environment measured by the Home Observation for Measurement of the Environment
Maternal parenting stress | 3 months of the child's age
  Maternal parenting stress measured by the Parenting Stress Index (PSI)
Child development | After child birth up to 3 months of the child's age
  Child developmental milestones measured by in-app questions
Child developmental milestones | 3 months of the child's age
  Child developmental milestones measured by the Survey of Well-being of Young Children (SWYC)

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Fatori, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No